CLINICAL TRIAL: NCT07164846
Title: Effect of Neuro20 Functional Electrical Stimulation Suit on Autonomic Function, Muscle Performance, and Gait
Acronym: Neuro20
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brooks Rehabilitation (Other)
Responsible Party: Principal Investigator, mark.bowden, Vice President of Clinical Integration and Research, Brooks Rehabilitation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00083882
Record Dates: First submitted 2025-08-07; First posted 2025-09-10 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Spinal Cord Injury; Stroke; Amputees
MeSH Terms: conditions — Spinal Cord Injuries; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Active Suit Stimulation (Experimental): Participants will be engaging in one hour of therapy with the suit in stimulation mode for twelve sessions. The first three sessions will be in conditioning mode, and the subsequent nine will be in strength mode.
  Interventions: Device: Therapy Sessions

INTERVENTIONS:
Device: Therapy Sessions — You will complete up to 12 sessions using the Neuro20 suit under the direct supervision of study staff. Each session will be 1-2 hours in duration. Each session, you will change into the suit and then receive no more than 105 minutes of electrical stimulation, and then change out of the suit and have a skin check. The suit has 20 electrodes that will stimulate muscles in your upper arm (above the elbow), upper leg (above the knee), chest, abdominals, and back. Stimulation levels will be adjusted to your comfort. You will likely feel tingling and/or muscle contractions. The timing and intensity of each type of activity will depend on your individual needs and will be prescribed by the study doctor.

SUMMARY:
This research aims to understand the effect of the Neuro20 Functional Electrical Stimulation Suit on autonomic nervous system function, muscle performance, and gait after amputation or neurologic injury.

DETAILED DESCRIPTION:
The purpose of this research study is to study the effect of the Neuro20 Functional Electrical Stimulation Suit on autonomic function, muscle performance, and walking ability. Electrical stimulation is intended to stimulate muscles in order to improve muscle performance. The Neuro20 is approved for this use by the United States Food and Drug Administration. In this study, the use of the device is considered investigational. Twenty subjects will participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* At least one week post amputation or neurologic injury (i.e. brain injury, stroke, spinal cord injury) and deemed medically stable to participate in rehabilitation
* Able to provide Informed Consent by demonstrating the ability to follow a three step command

Exclusion Criteria:

* Pacemaker / Defibrillator or severe cardiac disease (Class IV according to New York Heart Association Functional Classification)
* Implanted medical devices
* Active DVT/thrombophlebitis
* Active Cancer
* Active fever, infection, or acute inflammation
* Pregnancy
* Epilepsy or uncontrolled seizures or seizure within the last 6 months
* Implanted stimulator or pump that cannot be turned off externally
* Significant, active wounds in areas stimulated by the suit
* Inability to follow a three-step motor command
* Bleeding tendency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in Gait | Pre-intervention, mid-intervention at 1 week, and post-intervention at 4 weeks
  The 6-minute walk test is a simple, standardized test used to assess a person's exercise capacity and functional mobility. An increase in distance walked reflects an improvement in mobility and gait.

SECONDARY OUTCOMES:
Change in Autonomic Function | Pre-intervention, mid-intervention at 1 week, and post-intervention at 4 weeks
  Heart rate variability measures the variation in time between individual heartbeats, not just the average heart rate. An increase in variabiility indicates better health.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Bowden, PT, PhD, Principal Investigator — Brooks Rehabilitation
Locations (2):
- United States (2):
  - Brooks Rehabilitation, Jacksonville, Florida
  - The International Institute of Orthotics and Prosthetics, Tampa, Florida